CLINICAL TRIAL: NCT07286058
Title: A Phase 3, Multicenter, Long-Term Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of Zasocitinib (TAK-279) in Subjects With Active Psoriatic Arthritis Who Are Either Biologic DMARD-Naïve or Biologic DMARD-Experienced, Including Those With Inadequate Response to Biologic DMARDs
Brief Title: Continuation Study of Zasocitinib in Adults With Psoriatic Arthritis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-279-PsA-3003; 2025-522586-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-11; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Psoriatic Arthritis
Keywords: Drug Therapy; Latitude PsA; Latitude PsA-3003
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zasocitinib Dose A or Dose B (Experimental): Participants assigned to zasocitinib in the either parent studies (TAK-279-PsA-3001 [NCT06671483] or TAK-279-PsA-3002 [NCT06671496]) will continue to receive zasocitinib Dose A or Dose B at the same dose, oral tablets, QD for up to Week 104.
  Interventions: Drug: Zasocitinib
- Re-randomized Participants - Zasocitinib Dose A or Dose B (Experimental): Participants assigned to active comparator in the parent study (TAK-279-PsA-3001 [NCT06671483]) will be re-randomized to blinded treatment with zasocitinib Dose A or Dose B, oral tablets, QD for up to Week 104.
  Interventions: Drug: Zasocitinib

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib oral tablets.
  Other Names: TAK- 279; NDI-034858

SUMMARY:
Psoriatic arthritis (PsA) is a long-term inflammatory disease that affects the joints and skin.

The purpose of this study is to check how safe zasocitinib is, how well it is tolerated and how well it works in adults with PsA over a longer period of time.

Adults who completed the 1-year (52-week) treatment period in one of the parent studies (TAK-279-PsA-3001 [NCT06671483] or TAK-279-PsA-3002 [NCT06671496]) may be able to join this continuation study (also called long-term extension or LTE study). All participants in this continuation study, will receive zasocitinib (lower or higher dose), once a day (QD).

Each participant can be in this study for approximately 2 years (108 weeks). This includes a treatment period of up to 2 years (104 weeks) and a 1-month (4-week) follow-up period to monitor a participant's health.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is aged 18 years or older at the time of signing the informed consent form (ICF). In South Korea, the age requirement for adult participants is >=19 years of age.
2. The participant has completed the 52-week treatment period in one of the parent studies (TAK-279-PsA-3001 or TAK-279-PsA-3002) independent of treatment assignment, and without meeting the criteria for permanent discontinuation of trial intervention defined in the parent studies.
3. The participant must be deemed by the investigator to benefit from continued or newly initiated (that is, for participants randomized to active comparator in parent study TAK-279-PsA-3001) zasocitinib therapy.

Exclusion Criteria:

1. Any participant who is deemed by the investigator to be not benefiting from the trial intervention based upon lack of improvement or worsening of their symptoms in the respective parent study.
2. Any participant who met the criteria for permanent discontinuation of trial intervention defined in the parent studies (TAK-279-PsA-3001 or TAK-279-PsA-3002).
3. The participant has developed any disease(s) that might confound the evaluations of benefit of zasocitinib therapy since enrollment in the respective parent study, including but not limited to rheumatoid arthritis, axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, Lyme disease, gout, or fibromyalgia.
4. The participant has developed evidence of a concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the study assessments, such as evidence of non-plaque PsO (erythrodermic, pustular, predominately guttate PsO, inverse, or drug-induced PsO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1182 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2029-12-18 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From start of study drug administration up to follow-up (up to Week 108)
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. TEAE is defined as any AE emerging or manifesting at or after the initiation of treatment in the LTE study with a trial intervention or medicinal product or any existing AE that worsens in either intensity or frequency following exposure to the trial intervention or medicinal product. SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event.
Number of Participants With Adverse Events of Special Interest (AESI) | From start of study drug administration up to follow-up (up to Week 108)
  An AESI is an adverse event of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator may be appropriate.
Number of Participants With Clinically Significant Changes in Vital Sign Values | From start of study drug administration up to follow-up (up to Week 108)
  Vital signs will include measurement of body temperature, respiratory rate, sitting blood pressure and pulse rate. Any clinically significant change in vital signs will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Clinical Laboratory Values | From start of study drug administration up to follow-up (up to Week 108)
  Laboratory parameters will include hematology, chemistry and urinalysis. Any clinically significant change in laboratory values will be determined at the investigator's discretion.

SECONDARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology (ACR20) Response at Weeks 24, 48, and 104 | At Weeks 24, 48, and 104
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite clinical outcome assessment (COA) measure that includes both clinician-reported outcome assessments (ClinROs) and patient-reported outcomes (PROs). An ACR20 response is defined as greater than or equal to (>=) 20 percentage (%) improvement from baseline in both swollen joint count 66 joints (SJC66) and tender joint count 68 joints (TJC68), and >=20% improvement from baseline in 3 of the following 5 assessments: Patient's global assessment (PtGA) of PsA pain; PtGA of PsA; physician's global assessment of disease activity (PGA) of PsA; participant's assessment of physical function as measured by health assessment questionnaire-disability index (HAQ-DI); high-sensitivity C-reactive protein (hsCRP).
Percentage of Participants Achieving ACR50 at Weeks 24, 48, and 104 | At Weeks 24, 48, and 104
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs) and PROs. An ACR50 response is defined as >=50% improvement from baseline in both SJC66 and TJC68, and >=50% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP.
Percentage of Participants Achieving ACR70 at Weeks 24, 48, and 104 | At Weeks 24, 48, and 104
  ACR responses are the numerical measurement of improvement in multiple disease assessment criteria. It is a composite COA measure that includes both ClinROs) and PROs. An ACR70 response is defined as >=70% improvement from baseline in both SJC66 and TJC68, and >=70% improvement from baseline in 3 of the following 5 assessments: PtGA of PsA pain; PtGA of PsA; PGA of PsA; participant's assessment of physical function as measured by HAQ-DI; hsCRP.
Percentage of Participants Achieving Minimal Disease Activity (MDA) Status at Weeks 24, 48, and 104 | At Weeks 24, 48, and 104
  The MDA is defined as a composite outcome measure of 7 ClinROs and PROs used in PsA. Participants are classified as achieving MDA if they fulfil 5 of 7 outcome measures: TJC68 less than or equal to (<=) 1, SJC66 <=1, psoriasis area and severity index (PASI) score <=1 or body surface area (BSA) affected by psoriasis (PsO) <=3%, PtGA of PsA Pain score <=15, PtGA of PsA score <=20, HAQ-DI <=0.5, and Leeds Enthesitis Index (LEI) <=1.
Percentage of Participants Achieving >=75 % Improvement From Baseline in PASI Score at Weeks 24, 48, and 104 | At Weeks 24, 48, and 104
  A PASI-75 response is defined as >=75% improvement in the PASI score from baseline. It is a ClinRO used to measure PsO severity, combining the percentage of surface area of skin affected with the severity of erythema, induration, and desquamation across four body regions: head, upper extremities, trunk, and lower extremities. Severity is scored on a 0-4 scale, with 0 indicating a complete lack of cutaneous involvement and 4 indicating the severest possible involvement. PASI scores range from 0 to 72, with <=3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/